CLINICAL TRIAL: NCT01984398
Title: A Double-Blind Crossover Study In Healthy Volunteers to Compare Two Formulations of Androxal
Brief Title: Comparison of Two Formulations of Androxal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZA-110
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Enclomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12.5 mg Androxal (formulations A and B) (Experimental): 12.5 mg Androxal formulation A and 12.5 mg Androxal formulation B, a single dose of each formulation
  Interventions: Drug: 12.5 mg Androxal Formulation A; Drug: 12.5 mg Androxal Formulation B
- 25 mg Androxal (formulations A and B) (Experimental): 25 mg Androxal formulation A and 12.5 mg Androxal formulation B, a single dose of each formulation
  Interventions: Drug: 25 mg Androxal Formulation A; Drug: 25 mg Androxal Formulation B

INTERVENTIONS:
Drug: 12.5 mg Androxal Formulation A — Single dose of 12.5 mg Androxal formulation A
  Other Names: enclomiphene citrate
  Arms: 12.5 mg Androxal (formulations A and B)
Drug: 12.5 mg Androxal Formulation B — Single dose of 12.5 mg Androxal Formulation B
  Other Names: enclomiphene citrate
  Arms: 12.5 mg Androxal (formulations A and B)
Drug: 25 mg Androxal Formulation A — Single dose of 25 mg Androxal formulation A
  Other Names: enclomiphene citrate
  Arms: 25 mg Androxal (formulations A and B)
Drug: 25 mg Androxal Formulation B — Single dose of 25 mg Androxal formulation B
  Other Names: enclomiphene citrate
  Arms: 25 mg Androxal (formulations A and B)

SUMMARY:
To determine and compare the pharmacokinetics (PK) of a single dose of each of two formulations Androxal

DETAILED DESCRIPTION:
To determine and compare the pharmacokinetics (PK) of a single dose of each of two formulations of 12.5 mg and 25 mg Androxal administered to healthy male volunteers, and to determine and compare the safety of a single dose each of two formulations of 12.5 mg and 25 mg Androxal administered to healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Speaks, reads, and understands English or Spanish and is willing and able to provide written informed consent on an Institutional Review Board (IRB)-approved form prior to the initiation of any study procedures;
* Male, between the ages of 18-60 years;
* No significant abnormal findings at the screening physical examination as evaluated by the Investigator;
* Normal laboratory values (or abnormal but not clinically significant) at screening as determined by the Investigator;
* Subject is willing to remain in the clinic overnight for the Day 1 and Day 6 visits;
* Must be able to swallow gelatin capsules

Exclusion Criteria:

* Known hypersensitivity to Clomid;
* Abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Investigator;
* Subject with a significant organ abnormality or disease as determined by the Investigator;
* Any medical condition that would interfere with the study as determined by the Investigator;
* Slow Cytochrome P4502D6 (CYP2D6) metabolizer
* Participation in a clinical trial with investigational medication within 30 days prior to study medication administration;
* An acute illness within 5 days of study medication administration;;
* A mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude, as determined by the Investigator;
* History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism);
* History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia, or known history of (corrected QT) QTc interval prolongation;
* An employee or family member of an employee of the study site or the Sponsor.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (1):
- Clinical Pharmacology of miami, Miami, Florida, United States

REFERENCES:
- See also: Sponsor Corporate Website — http://www.reprosrx.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 12.5 mg Androxal (Formulation A), Then B; 12.5 mg Androxal (Formulation B), Then A: During Treatment Period 1, participants were randomly assigned to a single dose of either 12.5 mg Androxal Formulation A or 12.5 mg Androxal Formulation B.
  After the washout period, participants then crossed over to receive the alternate 12.5 mg formulation during Treatment Period 2, ensuring all participants had received one dose of Formulation A and one dose of Formulation B.
- 25 mg Androxal (Formulation A), Then B; 25 mg Androxal (Formulation B), Then A: During Treatment Period 1, participants were randomly assigned to a single dose of either 25 mg Androxal formulation A or 25 mg Androxal formulation B.
  After the washout period, participants then crossed over to receive the alternate 25 mg formulation during Treatment Period 2, ensuring all participants had received one dose of Formulation A and one dose of Formulation B.
Period: Treatment Period 1
Arm/Group | 12.5 mg Androxal (Formulation A), Then B | 12.5 mg Androxal (Formulation B), Then A | 25 mg Androxal (Formulation A), Then B | 25 mg Androxal (Formulation B), Then A
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of 5 to 7 Days
Arm/Group | 12.5 mg Androxal (Formulation A), Then B | 12.5 mg Androxal (Formulation B), Then A | 25 mg Androxal (Formulation A), Then B | 25 mg Androxal (Formulation B), Then A
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | 12.5 mg Androxal (Formulation A), Then B | 12.5 mg Androxal (Formulation B), Then A | 25 mg Androxal (Formulation A), Then B | 25 mg Androxal (Formulation B), Then A
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- 12.5 mg Androxal (Formulations A and B): During Treatment Period 1, participants were randomly assigned to a single dose of either 12.5 mg Androxal Formulation A or 12.5 mg Androxal Formulation B.
  After the washout period, participants then crossed over to receive the alternate 12.5 mg formulation during Treatment Period 2, ensuring all participants had received one dose of Formulation A and one dose of Formulation B.
- 25 mg Androxal (Formulations A and B): During Treatment Period 1, participants were randomly assigned to a single dose of either 25 mg Androxal formulation A or 25 mg Androxal formulation B.
  After the washout period, participants then crossed over to receive the alternate 25 mg formulation during Treatment Period 2, ensuring all participants had received one dose of Formulation A and one dose of Formulation B.
- Total: Total of all reporting groups
Arm/Group | 12.5 mg Androxal (Formulations A and B) | 25 mg Androxal (Formulations A and B) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (7.5) | 37.8 (6.1) | 37.7 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Androxal Cmax Formulation A
Description: To determine and compare the pharmacokinetic parameter Cmax between two formulations of Androxal
Time Frame: 24 hours
Population: Safety and PK populations are the same
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 12.5 mg Androxal Formulation A: A single dose of 12.5 mg Androxal formulation A, received either during Treatment Period 1 or Treatment Period 2.
- 25 mg Androxal Formulation A: A single dose of 25 mg Androxal Formulation A, received either during Treatment Period 1 or Treatment Period 2.
Arm/Group | 12.5 mg Androxal Formulation A | 25 mg Androxal Formulation A
Number analyzed (Participants) | 8 | 8
ng/mL | 0.999 (0.349) | 1.67 (0.74)

2. Primary Outcome: Androxal Cmax Formulation B
Description: To determine and compare the PK parameter Cmax between two formulations of Androxal
Time Frame: 24 hours
Population: Safety and PK populations are the same
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 12.5 mg Androxal Formulation B: A single dose of 12.5 mg Androxal formulation B, received either during Treatment Period 1 or Treatment Period 2.
- 25 mg Androxal Formulation B: A single dose of 25 mg Androxal formulation B, received either during Treatment Period 1 or Treatment Period 2.
Arm/Group | 12.5 mg Androxal Formulation B | 25 mg Androxal Formulation B
Number analyzed (Participants) | 8 | 8
ng/mL | 1.08 (0.42) | 1.74 (0.47)

ADVERSE EVENTS:
Time Frame: From Day 0 up to Day 8. (Up to 24 hours after last dose of study drug in Treatment Period 2)
Description: Adverse event data is presented for each Formulation (A and B) and dose (12.5mg and 25mg) of Androxal.
Groups:
- 12.5mg Androxal Formulation B: A single dose of 12.5 mg Androxal formulation B, received either during Treatment Period 1 or Treatment Period 2.
Arm/Group | 12.5 mg Androxal Formulation A | 12.5mg Androxal Formulation B | 25 mg Androxal Formulation A | 25 mg Androxal Formulation B
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 1/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12.5 mg Androxal Formulation A (N=8) | 12.5mg Androxal Formulation B (N=8) | 25 mg Androxal Formulation A (N=8) | 25 mg Androxal Formulation B (N=8)
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights